CLINICAL TRIAL: NCT00764257
Title: A Multicenter, Evaluator-Masked Study to Assess the Efficacy and Safety of Mentor's CX002 Dermal Filler Medical Device, When Applied as an Intradermal Implant for the Correction of Facial Wrinkles and Lip Augmentation (CX002 Dermal Filler Protocol)
Brief Title: PREVELLE Shape (CX002) Dermal Filler Protocol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mentor Worldwide, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 111990-0104-3
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Correction of Nasolabial Folds and Lip Augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PREVELLE Shape (Experimental)
  Interventions: Device: PREVELLE Shape
- Restylane (Active Comparator)
  Interventions: Device: Restylane

INTERVENTIONS:
Device: PREVELLE Shape
  Arms: PREVELLE Shape
Device: Restylane
  Arms: Restylane

SUMMARY:
The purpose of this study was to assess PREVELLE Shape (CX002), with respect to safety and efficacy for one year following treatment, for correction of facial nasolabial folds and when applied as an intradermal implant for lip augmentation.

ELIGIBILITY:
Inclusion Criteria

1. Subjects who gave written informed consent to participate.
2. Male or female subjects aged between 30 and 60 years inclusive (nasolabial fold cohort) or male or female subjects 18 years of age and older (lip augmentation cohort).
3. Subjects with NLFs that had shallow wrinkles, moderately deep wrinkles, or deep wrinkles with well defined edges (level 2, 3, or 4 on the six-point categorical rating scale), suitable for soft tissue augmentation or subjects who desired lip enlargement.

Exclusion Criteria

1. Subjects unwilling or unable to give written consent to participate in the investigation or unable to comply with the requirements of the protocol.
2. Subjects with a known hypersensitivity to sodium hyaluronate, lidocaine, xylocaine, or epinephrine.
3. Subjects with known severe allergies manifested by a history of anaphylaxis, or history or presence of severe multiple allergies.
4. Subjects with any serious skin disease, e.g., Eczema and psoriasis of the face, severe rosacea, scleroderma, local infections and severe acne.
5. Subjects with cancerous or precancerous lesions in either the right or left NLF or the lips.
6. Subjects with diabetes, coagulation disorders, connective tissue disorders, lipodystrophy, or other serious systemic disease.
7. Subjects with active herpes labialis.
8. Subjects infected with HIV and/or who received immunosuppressive therapy.
9. Subjects who received injections of resorbable tissue augmentation materials to the NLFs or the lips within 18 months prior to baseline.
10. Subjects who received permanent tissue implant materials to the NLFs or the lips.
11. Subjects who received any experimental drug or device within the previous three months.
12. Subjects who were to undergo another facial aesthetic procedure (including surgical, dermal implantation, Botox treatment, dermabrasion, facial massage, photo-aging treatments e.g., Retin-A and other related creams), during the entire 12-month study period
13. Subjects who were to undergo major facial plastic surgery (e.g. rhinoplasty with or without implant, eyelid lift, facelift, etc).
14. Subjects who were known alcohol or drug abusers.
15. Female subjects who were pregnant or lactating or were intending to become pregnant during the period of the study, or who would not use an adequate method of contraception (contraceptive pill, intra-uterine device) for the duration of the study.
16. Possessed any psychological condition, or was under treatment for any condition which, in the opinion of the Investigator and/or consulting physicians(s), would constitute an unwarranted risk.
17. Worked for Mentor or the study Investigator or were directly-related to anyone that worked for Mentor or the study doctor.
18. Subjects requiring facial soft tissue augmentation because of traumatic injury (nasolabial fold cohort only).
19. Subjects with none, just perceptible or very deep nasolabial wrinkles (0, 1, or, 5 points on the six-point Lemperle rating scale) (nasolabial fold cohort only).
20. Subjects who were treated with Retin-A four weeks prior to the baseline visit (nasolabial fold cohort only).
21. Subjects who were treated with Botox anywhere on the face within six months prior to the baseline visit (nasolabial fold cohort only).
22. Subjects who received laser resurfacing anywhere on the face within 12 months prior to the baseline visit (nasolabial fold cohort only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2004-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Study the safety and efficacy of CX002 when applied to the NLFs or lips. | 1 year
  The primary aim of the study is to assess CX002, with respect to safety and efficacy during the six months following treatment, in two subject cohorts:
  1. When applied as an intradermal implant for the correction of facial nasolabial folds (Nasolabial Fold Cohort). Nasolabial folds were chosen as the fold/wrinkle for treatment as they are often the most severe facial wrinkles, representing a "worst-case" scenario
  2. When applied as an intradermal implant for lip augmentation (Lip Augmentation Cohort)

CONTACTS AND LOCATIONS:
Locations (1):
- Mentor Worldwide, LLC, Santa Barbara, California, United States